CLINICAL TRIAL: NCT05884684
Title: What is the Potential Impact of Reviewing Post-procedure Images With Patients Following Interventional Spine Procedures.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, David Kohns, Principal Investigator, University of Michigan
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00216837
Record Dates: First submitted 2023-05-12; First posted 2023-06-01 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Patient Satisfaction
Keywords: Epidural; Spine procedure
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: A spine physician will not discuss images with the first group of participants immediately following their procedure. A spine physician will discuss images with the second group of participants immediately following their procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Post-Procedural Images Not Discussed with Participants (No Intervention): During a lumbar epidural steroid injection under fluoroscopic guidance, images are taken as part of the procedure. Following the procedure, the surgeon who performed it will not discuss the images with the participants in this arm.
  If participants request an explanation of the images, they will not be included in the analysis.
- Post-Procedural Images Discussed with Participants (Other): During a lumbar epidural steroid injection under fluoroscopic guidance, images are taken as part of the procedure. Following the procedure, the surgeon who performed it will discuss the images with the participants in this arm.
  Interventions: Other: Reviewing Imaging with Participant

INTERVENTIONS:
Other: Reviewing Imaging with Participant — Post-operatively, the images taken during the procedure will be reviewed with the participant.
  Arms: Post-Procedural Images Discussed with Participants

SUMMARY:
The purpose of this study is to explore the impact of spine physicians reviewing post-procedural fluoroscopic images with patients. The outcome measure to be assessed will be the potential impact the patient satisfaction and the patient's global impression of change (PGIC) 2 weeks after the spine procedure.

ELIGIBILITY:
Inclusion Criteria:

* Lumbosacral radiculopathy symptoms
* Received transforaminal epidural steroid injection

Exclusion Criteria:

* Patients who will be sedated for transforaminal epidural steroid injection
* Unable to read or understand English-language survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Modified Press Gainey Satisfaction (PGS) Questionnaire | Up to 2 hours following procedure in the post-op area
  Patient satisfaction as measured by a modified version of the PGS Questionnaire. The questionnaire is comprised of 9 questions measuring general patient satisfaction with the care experience. Each question is on a scale of 1 (very poor) to 5 (very good). The lowest possible score of the PGS is 9, and the highest possible score is 45. The lower the total score, the poorer the patient's satisfaction, while the higher the score, the higher the patient's satisfaction.

SECONDARY OUTCOMES:
Patient Global Impression of Change (PGIC) | 2 weeks following procedure
  The PGIC is a scale participants use to rate the level of change they have experienced following treatment. The PGIC is a 7-point scale from 1 (very much better) to 7 (very much worse). After making this selection, participants then rate the percentage of how their condition is following the transforaminal epidural steroid injection compared to before, with 10% being "a little better" and 100% being "very much better."

CONTACTS AND LOCATIONS:
Overall Officials: David Kohns, DO, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan - Burlington Building, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choudhury T, Jung J, Barnes M, Chandran S, Eckner JT, Geisser M, Kohns DJ. The impact on fluoroscopic image review on perceived benefit, patient satisfaction, and short-term improvement following lumbosacral epidural steroid injections. Interv Pain Med. 2025 Aug 31;4(3):100640. doi: 10.1016/j.inpm.2025.100640. eCollection 2025 Sep. PMID 40937359